CLINICAL TRIAL: NCT06370663
Title: A Single-arm, Exploratory Phase II Clinical Trial of Combined Radiotherapy and HAIC as First-line Treatment for Unresectable Locally Advanced Distal Cholangiocarcinoma
Brief Title: First-line Treatment for Unresectable Locally Advanced Distal Cholangiocarcinoma Combining Radiotherapy and HAIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to unacceptable treatment-related toxicity that raised safety concerns and outweighed the potential benefits.
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2023-109-01
Record Dates: First submitted 2024-04-06; First posted 2024-04-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic Cholangiocarcinoma; Radiotherapy; Hepatic Arterial Infusion Chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiotherapy; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Combining radiotherapy with Hepatic Arterial Infusion Chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy plus HAIC (Experimental): Radiotherapy + Hepatic Arterial Infusion Chemotherapy (Gesitabine) + Chemotherapy (GEMOX)
  Interventions: Radiation: Radiotherapy; Drug: HAIC (GEMOX); Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy + Hepatic Arterial Infusion Chemotherapy (Gesitabine) + Chemotherapy (GEMOX)
  Other Names: Hepatic Arterial Infusion Chemotherapy (GEMOX); Chemotherapy (Gesitabine)
Drug: HAIC (GEMOX) — Hepatic Arterial Infusion Chemotherapy (GEMOX)
  Other Names: HAIC
Drug: Chemotherapy — Chemotherapy (Gesitabine)
  Other Names: Chemotherapy (Gesitabine)

SUMMARY:
The median survival of intrahepatic cholangiocarcinoma remains less than one year, highlighting the need for new treatments. Hepatic arterial infusion chemotherapy (HAIC), especially with fluoropyrimidine-based regimens, has shown promise in ICC treatment due to increased local drug concentration and reduced systemic toxicity. A combined approach of radiotherapy and HAIC with gemcitabine infusion may offer a hopeful strategy for locally advanced cholangiocarcinoma. However, clinical research on this combination is lacking as first-line therapy for unresectable ICC. Therefore, a single-center, single-arm study aims to assess this treatment approach's safety, efficacy, and molecular predictors. Improved HAIC delivery through modified percutaneous implantation provides a reliable pathway for effective treatment. In conclusion, exploring the synergistic effects of radiotherapy and HAIC in ICC could pave the way for more effective and personalized treatment strategies for this challenging cancer type.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) ranks as the second most common primary liver cancer, constituting 15%-20% of malignant liver tumors, with a rising incidence trend. Unlike hepatocellular carcinoma (HCC), ICC displays higher invasiveness and metastatic potential. Surgical resection remains the optimal treatment, yet many patients present with unresectable disease or metastasis, limiting surgical options. Chemotherapy, particularly the GC regimen, is standard for unresectable and metastatic ICC. Studies like ABC-02 have improved survival with GC chemotherapy compared to gemcitabine monotherapy. However, the median survival remains less than one year, highlighting the need for new treatments. Hepatic arterial infusion chemotherapy (HAIC), especially with fluoropyrimidine-based regimens, has shown promise in ICC treatment due to increased local drug concentration and reduced systemic toxicity. A combined approach of radiotherapy and HAIC with gemcitabine infusion may offer a hopeful strategy for locally advanced cholangiocarcinoma. However, clinical research on this combination is lacking as first-line therapy for unresectable ICC. Therefore, a single-center, single-arm study aims to assess this treatment approach's safety, efficacy, and molecular predictors. Improved HAIC delivery through modified percutaneous implantation provides a reliable pathway for effective treatment. In conclusion, exploring the synergistic effects of radiotherapy and HAIC in ICC could pave the way for more effective and personalized treatment strategies for this challenging cancer type.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, both male and female.
* Histologically or cytologically confirmed primary cholangiocarcinoma (including intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, and gallbladder carcinoma) or imaging-confirmed localized cholangiocarcinoma, staged as T1-4N0/N+M0 (according to AJCC 7th edition clinical staging).
* Ineligible for surgical treatment or refusal of surgical treatment upon pre-treatment assessment.
* Presence of measurable lesions as per RECIST v1.1 criteria for evaluation.
* ECOG performance status: 0-1.
* Expected survival of more than 6 months.
* Tolerable function of major organs for treatment.
* Non-surgically sterilized or premenopausal female patients need to use a medically accepted contraceptive method during the study treatment period and within 3 months after the end of the study treatment.

Exclusion Criteria:

* Subjects with any active autoimmune disease or a history of autoimmune disease are excluded.
* Patients with poorly controlled clinical symptoms or diseases related to the heart, such as:

  1. NYHA Class 2 or above heart failure
  2. Unstable angina
  3. Myocardial infarction within the past year
  4. Clinically significant ventricular or supraventricular arrhythmias requiring treatment or intervention
  5. QTc >450 ms (males); QTc >470 ms (females)
* Abnormal coagulation function (INR >1.5 or PT >16s), bleeding tendencies, or receiving thrombolytic or anticoagulant therapy.
* Subjects who have received radiation therapy, chemotherapy, steroid therapy, surgery, or molecular targeted therapy within less than 4 weeks (or 5 half-lives of the drug, whichever is longer) before the study drug's first dose, or who have not recovered from adverse events caused by previous treatment (excluding alopecia) to ≤Grade 1 according to CTCAE.
* Subjects with clinically symptomatic ascites, pleural effusion, or pericardial effusion requiring therapeutic puncture or drainage. Those who have had stable ascites or effusion after drainage of pleural or pericardial effusion for at least 2 weeks before the first dose of the study drug can be included in the study.
* Subjects with significant hemoptysis in the last 2 months or hemoptysis of half a teaspoon (2.5 ml) or more.
* Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophiliacs, coagulation disorders, thrombocytopenia, splenomegaly, etc.) or those who have had arterial or venous thrombotic events within the last 6 months (prior to first SHR-1210 administration).
* Subjects with active infections or unexplained fever >38.5°C during screening or before the first dose of the study drug.
* Patients with objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe lung function impairment, etc., either historically or currently.
* Subjects with congenital or acquired immunodeficiency (such as HIV infection) or active hepatitis (HBV reference: HBV DNA test value exceeds the upper limit of normal; HCV reference: HCV virus titer or RNA test value exceeds the upper limit of normal).
* Use of other investigational drugs within 4 weeks prior to the first dose of the study drug.
* Subjects with a history of or concurrent other malignancies (excluding cured basal cell carcinoma and cervical carcinoma in situ).
* Subjects who may receive other systemic anti-tumor therapies during the study.
* Subjects who have previously received PD-1 antibody therapy or immune therapy targeting PD-1/PD-L1.
* Vaccination with live vaccines within less than 4 weeks before the study drug's administration or potentially during the study period.
* Other factors judged by the investigator that may necessitate premature termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 2 year
  Assessing the severity of adverse events according to CTCAE v4.0.3 standards.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 year
  the length of time during and after treatment with a medication or therapy that a patient lives with the disease without it progressing

CONTACTS AND LOCATIONS:
Overall Officials: Jin Bo Yue, Dr., Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Jinbo Yue, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banales JM, Cardinale V, Carpino G, Marzioni M, Andersen JB, Invernizzi P, Lind GE, Folseraas T, Forbes SJ, Fouassier L, Geier A, Calvisi DF, Mertens JC, Trauner M, Benedetti A, Maroni L, Vaquero J, Macias RI, Raggi C, Perugorria MJ, Gaudio E, Boberg KM, Marin JJ, Alvaro D. Expert consensus document: Cholangiocarcinoma: current knowledge and future perspectives consensus statement from the European Network for the Study of Cholangiocarcinoma (ENS-CCA). Nat Rev Gastroenterol Hepatol. 2016 May;13(5):261-80. doi: 10.1038/nrgastro.2016.51. Epub 2016 Apr 20. PMID 27095655
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Fiteni F, Nguyen T, Vernerey D, Paillard MJ, Kim S, Demarchi M, Fein F, Borg C, Bonnetain F, Pivot X. Cisplatin/gemcitabine or oxaliplatin/gemcitabine in the treatment of advanced biliary tract cancer: a systematic review. Cancer Med. 2014 Dec;3(6):1502-11. doi: 10.1002/cam4.299. Epub 2014 Aug 11. PMID 25111859
- [Result] Kim ST, Kang JH, Lee J, Lee HW, Oh SY, Jang JS, Lee MA, Sohn BS, Yoon SY, Choi HJ, Hong JH, Kim MJ, Kim S, Park YS, Park JO, Lim HY. Capecitabine plus oxaliplatin versus gemcitabine plus oxaliplatin as first-line therapy for advanced biliary tract cancers: a multicenter, open-label, randomized, phase III, noninferiority trial. Ann Oncol. 2019 May 1;30(5):788-795. doi: 10.1093/annonc/mdz058. PMID 30785198
- [Result] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Result] Zhang J, Wu L, Liu J, Lin M. A metastatic intrahepatic cholangiocarcinoma treated with programmed cell death 1 inhibitor: a case report and literature review. Immunotherapy. 2020 Jun;12(8):555-561. doi: 10.2217/imt-2019-0100. Epub 2020 May 6. PMID 32372672
- [Result] Jarnagin WR, Schwartz LH, Gultekin DH, Gonen M, Haviland D, Shia J, D'Angelica M, Fong Y, DeMatteo R, Tse A, Blumgart LH, Kemeny N. Regional chemotherapy for unresectable primary liver cancer: results of a phase II clinical trial and assessment of DCE-MRI as a biomarker of survival. Ann Oncol. 2009 Sep;20(9):1589-1595. doi: 10.1093/annonc/mdp029. Epub 2009 Jun 2. PMID 19491285
- [Result] Konstantinidis IT, Groot Koerkamp B, Do RK, Gonen M, Fong Y, Allen PJ, D'Angelica MI, Kingham TP, DeMatteo RP, Klimstra DS, Kemeny NE, Jarnagin WR. Unresectable intrahepatic cholangiocarcinoma: Systemic plus hepatic arterial infusion chemotherapy is associated with longer survival in comparison with systemic chemotherapy alone. Cancer. 2016 Mar 1;122(5):758-65. doi: 10.1002/cncr.29824. Epub 2015 Dec 22. PMID 26695839